CLINICAL TRIAL: NCT00506233
Title: Feasibility Study of Collecting Multicenter Chronic GVHD Data
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2006-0541
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Graft-Versus-Host Disease
Keywords: Graft-Versus-Host Disease; GVHD; Questionnaire
MeSH Terms: conditions — Graft vs Host Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Chronic Graft-Versus Host Disease (GvHD): Participants with chronic graft-versus host disease (GvHD)
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Completion of questionnaires at 3 different times (when joining this study, 3 months later, and 6 months later). Each should take about 20-30 minutes to complete.
  Other Names: surveys

SUMMARY:
Primary Objective:

1. To determine the feasibility of conducting a multi-site longitudinal observational study of patients with chronic graft-versus-host disease (GVHD).

DETAILED DESCRIPTION:
If you agree to take part in this study, you will be asked to fill-out some questionnaires, and your medical records will be reviewed. Your doctor or healthcare provider will also be asked to complete a questionnaire.

You will be asked to fill-out questionnaires at 3 different times (when you join this study, 3 months later, and 6 months later). The questionnaires will include questions about how your chronic GvHD impacts your body, your day-to-day activities, your emotions and perceptions, and your social and sexual life. Each questionnaire has 195 questions. Each should take about 20-30 minutes to complete, but you will also be asked how long it takes you to complete each questionnaire. For most participants, these visits will be part of your routine schedule for follow-up for the disease.

You have several options for where you may choose to complete the questionnaires. They may be completed when you visit the doctor for your appointments, at home (you will have to mail them back in self-addressed stamped envelopes that will be provided to you), or over the internet. If you are interested in the internet option, please ask study staff for more details. If at any time, your healthcare provider does not think it would be in your best interest to receive a survey at one of your scheduled time points, you will not be given a survey at that time, and you will be taken off this study.

Your healthcare provider will be asked to fill-out a questionnaire that asks about what was found on your physical exam and routine laboratory tests, what medications you are taking, and how severe your chronic GvHD is at that clinic visit.

Your medical records will be reviewed for about 1 year after your enrollment in this study to collect information about your stem cell transplant procedure, your medications, your medical condition, and the results of tests and procedures. The reviewing of your medical records does not require your active participation.

You will be on this study until you have completed the 6-month questionnaire.

This is an investigational study. There is no cost involved for participation in this study. Up to 40 participants will take part in this multicenter study. Up to 15 will be enrolled M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 2 years
2. Prior allogeneic stem cell transplant, with any graft source, donor type, and GVHD prophylaxis allowed
3. If a prevalent case (defined as enrollment three or more months after chronic GVHD diagnosis), then subject must be within 2 years of stem cell infusion
4. Diagnosis of chronic GVHD meeting the diagnostic criteria of the diagnosis and staging group of the NIH consensus conference
5. Need for systemic treatment, defined as any medication or intervention delivered systemically, including extracorporeal photopheresis. If a patient only received topical or local therapy at diagnosis, but subsequently requires systemic treatment, they may be enrolled upon initiation of systemic therapy. (Note, these patients will be classified as incident or prevalent cases depending on time from chronic GVHD diagnosis, not start of systemic therapy)
6. Progression-free for their malignancy at enrollment (no evidence of primary disease progression since transplant, although residual disease may still be present)
7. Evaluation at the transplant center at the time of study enrollment, and agreement to be re-evaluated at the transplant center at 3 and 6 months
8. Signed, informed consent and if applicable, child assent

Exclusion Criteria:

1. Inability to verbally communicate in English
2. Inability to comply with study procedures
3. Anticipated survival less than 6 months due to co-morbid disease or persistent malignancy

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants with chronic graft-versus host disease (GvHD) at UT MD Anderson Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2006-08; Primary Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amin Alousi, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - U.T.M.D. Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org